CLINICAL TRIAL: NCT01450566
Title: Intraureteral of Alkalinized Lidocaine as Novel Approach to Post-Ureteroscopy Pain: Double-blind Prospective Randomized Controlled Trial
Brief Title: Intraureteral Lidocaine for Post-Ureteroscopy Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Darren Beiko, Principal Investigator and Associate Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Lidocaine Beiko
Record Dates: First submitted 2011-09-20; First posted 2011-10-12 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Ureteral Calculi; Renal Calculi
Keywords: ureteroscopy (URS); ureteral stent placement; Ureteral Calculi; Renal Calculi
MeSH Terms: conditions — Ureteral Calculi; Kidney Calculi | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Experimental): Use of lidocaine
  Interventions: Drug: Lidocaine
- No lidocaine (Placebo Comparator): No lidocaine/standard of care
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine — Use of lidocaine
  Arms: Lidocaine
Drug: Saline — Saline
  Arms: No lidocaine

SUMMARY:
Ureteroscopy (URS) is minimally invasive procedure for management of renal stones. URS is often involves concomitant of an indwelling ureteral stents. Placements of these stents include pain, bladder irritability, infection, migration, encrustation and stones.

Pain is one of most significant problem of ureteral stents. There are no satisfactory measures to deal with this problem. A novel approach to manage the pain is to load a drug onto ureteral stent and deliver the drug into the urinary tract at controlled release rate.

Lidocaine has been proven to be effective for management of the pain associated with interstitial cystitis. This agent has the potential for management of post-URS pain.

DETAILED DESCRIPTION:
Patients treated with ureteroscopy (URS) for ureteral or renal calculi requiring a ureteral stent at time of URS will be randomized to receive intraureteral instillation of alkalinized lidocaine hydrochloride (study group) or normal saline (control group) immediately following the procedure to assess safety and effectiveness in alleviating pain and stent symptoms. Thousands of removable stents are placed in patients' ureters (tubes connecting kidney and bladder) each year in Canada. These plastic stents allow the kidney to drain when there is swelling after kidney stone surgery or if they are otherwise obstructed. Studies report that more than 80% of patients have painful symptoms from indwelling ureteral stents. This study will attempt to show that local anesthetic injected directly into the ureter before stent placement will reduce stent pain. Recent studies have shown infusing lidocaine with bicarbonate (a local anesthetic) into painful bladders is safe, and patients' symptoms improve dramatically. This result inspired the innovative idea that injecting a similar solution into the kidney and ureter (which have the same lining as the bladder) will numb the area sufficiently to decrease stent related pain.

The study will randomly select half of the patients to receive an injection of non-irritating salt water (placebo), and half an injection of pH buffered lidocaine before the stent is placed. Both patients and physicians will be blinded to the assignment of treatment or placebo. The investigators will then compare pain scores post operatively.

If successful, future researchers may use lidocaine in drug eluding stents to further ameliorate pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing URS for treatment of a urinary calculus who requires placement of ureteral stent on a string
* Able to undergo a general anaesthetic
* At least 18 years old
* Willing and able to complete patient symptom questionnaires

Exclusion Criteria:

* Solitary Kidney
* Renal failure
* Anatomic bladder or ureteral abnormality
* Uncorrected coagulopathy
* Previous cystectomy or urinary diversion
* Neurogenic bladder
* Interstitial cystitis
* Transplanted kidney
* Pregnancy
* Requires an indwelling catheter
* Recurrent urinary tract infections
* Requires an indwelling stent
* Pelvic kidney
* Requires bilateral treatment/stents
* Previous bladder or ureteral reconstructive surgery
* Ureteral perforation during procedure
* Ureteral stenting, within one month of URS
* Known sensitivity to lidocaine
* Febrile at time of randomization or treatment
* Requires spinal anaesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Pain as measured by the mean VAS pain score over the study period. | 7 days
  Pain as measured by the mean VAS pain score over the study period. VAS pain, urinary frequency, pain mediation diary and ureteral stent symptoms assessed at different time points during the study. Efficacy will be determined by a 2 or more point mean difference in pain scores between the active treatment group and placebo group.

SECONDARY OUTCOMES:
Establishment of safety of intraureteral administration of the alkalinized lidocaine solution | 7 days
  Comparison of safety parameters (adverse events) between placebo and treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Darren Beiko, MD FRCSC, Principal Investigator — Queen's University
Locations (1):
- Centre for Applied Urological Research/Kingston General Hospital, Kingston, Ontario, Canada